CLINICAL TRIAL: NCT05625061
Title: A Micro-randomized Trial of JITAI Messaging to Improve Adherence to Multiple Weight Loss Behaviors in Young Adults
Brief Title: Just-in-time Adaptive Intervention Messaging in a Digital Weight Loss Intervention for Young Adults
Acronym: Nudge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 22-0170; 1R01HL161373 (NIH)
Record Dates: First submitted 2022-11-14; First posted 2022-11-22 (Actual); Results first posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-01

CONDITIONS: Obesity; Overweight; Overweight and Obesity
Keywords: Mobile intervention; Diet; Physical Activity; Behavioral weight loss
MeSH Terms: conditions — Obesity; Overweight; Motor Activity | interventions — Methods

STUDY DESIGN:
Intervention Model Description: This is a micro-randomized trial, a form of a sequential, factorial trial. At every time point, a participant is micro-randomized to receive or not receive an intervention message.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Core Behavioral Weight Loss (BWL) Intervention (Experimental): Behavioral weight loss core intervention, includes activity tracker, wireless scale, daily self-weighing, and smartphone app with weekly behavioral lessons, food tracking log, weekly tailored feedback summary, and daily weight-related behavioral goals. Core intervention component is combined with each of the 7 intervention messages to be tested repeatedly over time.
  Interventions: Behavioral: Core Behavioral Weight Loss (BWL) Intervention
- Core BWL Intervention + BCT 1 Message (Action Planning) (Experimental): Core BWL Intervention + Message testing the Behavior Change Technique "Action Planning"
  Interventions: Behavioral: Behavior Change Technique 1 Message (Action Planning)
- Core BWL Intervention + BCT 2 Message (Discrepancy) (Experimental): Core BWL Intervention + Message testing the Behavior Change Technique "Discrepancy Between Current Behavior and Goal"
  Interventions: Behavioral: Behavior Change Technique 2 Message (Discrepancy between Current Behavior and Goal)
- Core BWL Intervention + BCT 3 Message (Feedback on Outcome of Behavior) (Experimental): Core BWL Intervention + Message testing the Behavior Change Technique "Feedback on Outcome of Behavior"
  Interventions: Behavioral: Behavior Change Technique 3 Message (Feedback on Outcome of Behavior)
- Core BWL Intervention + BCT 4 Message (Social Support) (Experimental): Core BWL Intervention + Message testing the Behavior Change Technique "Social Support"
  Interventions: Behavioral: Behavior Change Technique 4 Message (Social Support)
- Core BWL Intervention + BCT 5 Message (Social Comparison) (Experimental): Core BWL Intervention + Message testing the Behavior Change Technique "Social Comparison"
  Interventions: Behavioral: Behavior Change Technique 5 Message (Social Comparison)
- Core BWL Intervention + BCT 6 Message (Social Reward) (Experimental): Core BWL Intervention + Message testing the Behavior Change Technique "Social Reward"
  Interventions: Behavioral: Behavior Change Technique 6 Message (Social Reward)
- Core BWL Intervention + BCT 7 Message (Focus on Past Success) (Experimental): Core BWL Intervention + Message testing the Behavior Change Technique "Focus on Past Success"
  Interventions: Behavioral: Behavior Change Technique 7 Message (Focus on Past Success)

INTERVENTIONS:
Behavioral: Core Behavioral Weight Loss (BWL) Intervention — All participants receive a mobile behavioral weight loss intervention delivered through a study smartphone app with weekly behavioral lessons, food tracking log, weekly tailored feedback, and daily weight-related behavioral goals; a connected physical activity tracker and wireless scale. As micro-randomized trials are sequential, full factorial experiments, this core intervention component is combined with each of the 7 intervention messages (i.e., Behavior Change Technique (BCT) messages) to be tested repeatedly over time.
  Participants will be evaluated at each of 3 decision points (morning, midday, evening) on each day of the study, and if eligible then micro-randomized, to receive or not receive, 1 of 7 types of daily intervention messages promoting achievement of proximal weight-related behavioral goals.
  Arms: Core Behavioral Weight Loss (BWL) Intervention
Behavioral: Behavior Change Technique 1 Message (Action Planning) — Core BWL Intervention + Message in smartphone app prompts detailed planning of performance of one of the 3 target behaviors (daily weighing, active minutes, red food intake).
  Arms: Core BWL Intervention + BCT 1 Message (Action Planning)
Behavioral: Behavior Change Technique 2 Message (Discrepancy between Current Behavior and Goal) — Core BWL Intervention + Message in smartphone app provides feedback on each of the 3 target behaviors (daily weighing, active minutes, red food intake) in the form of information drawing attention to discrepancies between participants' current behavior and participants' daily goals.
  Arms: Core BWL Intervention + BCT 2 Message (Discrepancy)
Behavioral: Behavior Change Technique 3 Message (Feedback on Outcome of Behavior) — Core BWL Intervention + Message in smartphone app provides participants with feedback on their weight change, relating it to their performance on one of the 3 target behaviors (daily weighing, active minutes, red food intake).
  Arms: Core BWL Intervention + BCT 3 Message (Feedback on Outcome of Behavior)
Behavioral: Behavior Change Technique 4 Message (Social Support) — Core BWL Intervention + Message in smartphone app advises participants on eliciting the provision of social support from their existing network related to one of the 3 target behaviors (daily weighing, active minutes, red food intake).
  Arms: Core BWL Intervention + BCT 4 Message (Social Support)
Behavioral: Behavior Change Technique 5 Message (Social Comparison) — Core BWL Intervention + Message in smartphone app systematically induces comparison of participants' behavioral performance with other participants, including general, upward (i.e., comparison to participants doing better: weighing more, engaging in more activity, staying within red food limits), and downward comparisons (to participants doing worse).
  Arms: Core BWL Intervention + BCT 5 Message (Social Comparison)
Behavioral: Behavior Change Technique 6 Message (Social Reward) — Core BWL Intervention + Message in smartphone app reinforces participants' effort or progress in performing one of the 3 target behaviors (daily weighing, active minutes, red food intake).
  Arms: Core BWL Intervention + BCT 6 Message (Social Reward)
Behavioral: Behavior Change Technique 7 Message (Focus on Past Success) — Core BWL Intervention + Message in smartphone app advises participants to think about or list previous successes related to performing one of the 3 target behaviors (daily weighing, active minutes, red food intake).
  Arms: Core BWL Intervention + BCT 7 Message (Focus on Past Success)

SUMMARY:
The purpose of this micro-randomized trial is to evaluate the effects of 7 types of intervention messages targeting specific behavior change techniques (i.e., BCT messages) delivered in "just-in-time" (JIT) moments on daily achievement of weight-related behavioral goals among n=201 young adults with overweight and obesity, participating in a digital, mobile comprehensive lifestyle intervention. "Just-in-time adaptive interventions" (JITAIs) are an alternative to the "one size fits all" approach of mobile intervention development that can provide tailored, real-time messaging and support for young adults.

DETAILED DESCRIPTION:
An estimated 1 in 2 US adults will have obesity by 2030, which is a major cause of morbidity and mortality. The highest risk of weight gain is among young adults ages 18-35 years. In-person behavioral interventions generally produce clinically significant weight losses, but cost and reduced reach limit their ability to impact obesity at a population level. Web-based interventions that mimic the structure of weekly face-to-face treatment have proven a viable alternative, though weight losses are generally smaller than in-person treatment. Mobile treatments have the potential for high reach, but have been less effective, producing 1-3 kgs over 6 months. Newer digital intervention approaches called "just-in-time adaptive interventions" (JITAIs) promise to improve upon mobile outcomes by offering adaptive, personalized feedback on behavior, which consists of providing the "right type of support" at "the right time" rather than on a fixed schedule. This "just-in- time," or JIT, approach is made possible by the emergence of low-cost and widely available digital health tools that allow for the collection of continually updated health data. However, to date, no JITAIs have successfully targeted multiple weight-related behaviors (weighing, activity, and diet), and there has been no systematic examination of what types of messaging interventions best promote adherence to these three weight loss behaviors, for whom they are effective, and under what conditions. To address this problem, a micro-randomized trial will be used to evaluate the effects of 7 types of intervention messages targeting specific behavior change techniques (i.e., BCT messages) delivered in JIT moments on daily achievement of behavioral goals among n=201 young adults with overweight and obesity. All participants will receive a 6-month behavioral weight loss intervention using our Nudge mobile app, which includes evidence-based weekly lessons, tailored feedback, self-monitoring, and daily BCT messages. Participants will receive a wireless scale, activity tracker, and track "red" foods (high-calorie foods) in the app and have 3 goals: weigh daily, a daily active minutes goal that gradually increases if met, and a daily red foods limit. At 3 decision points per day, participants will be micro-randomized to receive or not receive 1 of 7 types of BCT messages. Each intervention message has unique decision rules for availability. Candidate intervention message options have been carefully selected from empirical evidence, tested in our prior studies, or are from our pilot micro-randomized trial. Assessments will occur daily, and at 0, 3 and 6 months, to accomplish the following specific aims: 1) Evaluate the effects of each behavior change technique message (i.e., BCT message) on daily adherence to weight loss behaviors; 2) Determine whether the effects of BCT messages on proximal outcomes change over time; and 3) Assess whether the effects of BCT messages on proximal outcomes are moderated by participants' contextual factors. Findings will guide how adaptive, behaviorally- and contextually-dependent messages are incorporated into future JITAIs for weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of 25 - 45 kg/m^2 at baseline
* English-speaking, reading, and writing
* Own a smartphone with a data and text messaging plan

Exclusion Criteria:

* Type 1 diabetes or currently receiving medical treatment for Type 2 diabetes
* Report a heart condition, chest pain during periods of activity or rest, or loss of consciousness on the Physical Activity Readiness Questionnaire (PAR-Q; items 1-4).
* Other health problems which may influence the ability to walk for physical activity or be associated with unintentional weight change, including cancer treatment within the past 5 years or tuberculosis
* Lost 10 lbs. or more of body weight (and kept it off) in the last 6 months
* Past diagnosis of or receiving treatment for a clinically diagnosed eating disorder (anorexia nervosa or bulimia nervosa)
* Current symptoms of alcohol or substance dependence
* Currently pregnant, pregnant within the past 6 months, or planning to become pregnant within the next 6 months
* Untreated thyroid disease or any changes (type or dose) in thyroid medication in last 6 months
* Hospitalization for depression or other psychiatric disorder within the past 12 months
* History of psychotic disorder or bipolar disorder
* Currently participating in a weight loss, nutrition, or physical activity study or program or other study that would interfere with this study
* Currently using prescription medications with known effects on appetite or weight (e.g., oral steroids, weight loss medications), with the exception of individuals on a stable dose of Selective Serotonin Reuptake Inhibitors (SSRIs) for 3 months)
* Previous surgical procedure for weight loss or planned weight loss surgery in the next year
* Another member of the household is a participant or staff member on this trial
* Reason to suspect that the participant would not adhere to the study intervention
* Reside outside of the United States
* Have participated in another study conducted by the UNC Weight Research Program within the past 12 months

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 255 (Actual)
Dates: Start 2023-08-25 (Actual); Primary Completion 2025-01-05 (Actual); Study Completion 2025-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carmina G. Valle, PhD, MPH, Principal Investigator — Assistant Professor
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 12 to 36 months following publication provided the investigator who proposes to use the data has submitted a written proposal to the Principal Investigator describing the intended use of the data and approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC. The release of specific data may be delayed if data are part of an analysis being prepared for a separate publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: beginning at 12 and continuing for 36 months following publication
Access Criteria: Investigator has UNC PI-approved proposal, institutional IRB, IEC, or REB approval and an executed data use/sharing agreement with UNC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 911 individuals completed the online screening survey; 533 met initial eligibility criteria; and 255 signed informed consent. Following consent, 206 completed all required onboarding and baseline measurement procedures and began the study.
Pre-assignment Details: Participants who signed informed consent were required to complete all onboarding steps, including baseline surveys, remote weight measurements, and the kickoff session. The 206 who completed these procedures and remained eligible began the study.
Period: Overall Study
Arm/Group | Core Behavioral Weight Loss (BWL) Intervention
Started | 206
Completed 3-Month Visit | 204
Completed | 201
Not Completed | 5
Not completed — Withdrawal by Subject | 4
Not completed — Intervention Suspended | 1

BASELINE CHARACTERISTICS:
Arm/Group | Core Behavioral Weight Loss (BWL) Intervention
Number analyzed (Participants) | 206
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.8 (5.5)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex (NIH/OMB): Female | 134
  Sex (NIH/OMB): Male | 71
  Sex (NIH/OMB): Prefer not to answer | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 20
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 20
  White | 148
  More than one race | 8
  Unknown or Not Reported | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34
  Not Hispanic or Latino | 169
  Unknown or Not Reported | 3
Weight (kg) [Mean (Standard Deviation); unit: kilograms] | 94.5 (20.1)

OUTCOME MEASURES:

1. Primary Outcome: Met Daily Weighing Goal
Description: Each observation corresponds to a microrandomization decision point; the reported value reflects the outcome measured within that unit. Among the randomization observations in which the participant had not yet weighed, this outcome is the number of observations in which the daily weighing goal was met after receiving or not receiving a message and before the end of the day. Observations are accumulated across participants and across time. On the day of randomization, a dichotomous outcome of whether a participant weighed or did not weigh is calculated.
Time Frame: Daily throughout the study, a total of up to 24 weeks
Population: The number of observations analyzed in each arm reflects the total number of observations (across participants, across the study) in which a message of that type was either received or not received, as noted in the arm description. The number of participants analyzed is the total number of participants whose observations are included in that particular arm. The Social Reward BCT was not delivered for the outcome of daily weighing and thus no data were collected for BCT 6.
Measure: Number; unit: goals met
Units Other Than Participants: Observations
Groups:
- Any Message: Received: All observations in which microrandomization resulted in receiving the message (a message with any behavior or BCT).
- Any Message: Not Received: All observations in which microrandomization resulted in not receiving the message (a message with any behavior or BCT).
- Weighing Message: Received: All observations in which weighing was the assigned behavior and microrandomization resulted in receiving the message (with any BCT).
- Weighing Message: Not Received: All observations in which weighing was the assigned behavior and microrandomization resulted in not receiving the message (with any BCT).
- Weighing BCT 1 Message (Action Planning): Received: All observations in which weighing was the assigned behavior, Action Planning was the selected BCT type, and microrandomization resulted in receiving the message.
- Weighing BCT 1 Message (Action Planning): Not Received: All observations in which weighing was the assigned behavior, Action Planning was the selected BCT type, and microrandomization resulted in not receiving the message.
- Weighing BCT 2 Message (Discrepancy): Received: All observations in which weighing was the assigned behavior, Discrepancy was the selected BCT type, and microrandomization resulted in receiving the message.
- Weighing BCT 2 Message (Discrepancy): Not Received: All observations in which weighing was the assigned behavior, Discrepancy was the selected BCT type, and microrandomization resulted in not receiving the message.
- Weighing BCT 3 Message (Feedback on Outcome of Behavior): Received: All observations in which weighing was the assigned behavior, Feedback on Outcome of Behavior was the selected BCT type, and microrandomization resulted in receiving the message.
- Weighing BCT 3 Message (Feedback on Outcome of Behavior): Not Received: All observations in which weighing was the assigned behavior, Feedback on Outcome of Behavior was the selected BCT type, and microrandomization resulted in not receiving the message.
- Weighing BCT 4 Message (Social Support): Received: All observations in which weighing was the assigned behavior, Social Support was the selected BCT type, and microrandomization resulted in receiving the message.
- Weighing BCT 4 Message (Social Support): Not Received: All observations in which weighing was the assigned behavior, Social Support was the selected BCT type, and microrandomization resulted in not receiving the message.
- Weighing BCT 5 Message (Social Comparison): Received: All observations in which weighing was the assigned behavior, Social Comparison was the selected BCT type, and microrandomization resulted in receiving the message.
- Weighing BCT 5 Message (Social Comparison): Not Received: All observations in which weighing was the assigned behavior, Social Comparison was the selected BCT type, and microrandomization resulted in not receiving the message.
- Weighing BCT 6 Message (Social Reward): Received: All observations in which weighing was the assigned behavior, Social Reward was the selected BCT type, and microrandomization resulted in receiving the message.
- Weighing BCT 6 (Social Reward) Message: Not Received: All observations in which weighing was the assigned behavior, Social Reward was the selected BCT type, and microrandomization resulted in not receiving the message.
- Weighing BCT 7 Message (Focus on Past Success): Received: All observations in which weighing was the assigned behavior, Focus on Past Success was the selected BCT type, and microrandomization resulted in receiving the message.
- Weighing BCT 7 Message (Focus on Past Success): Not Received: All observations in which weighing was the assigned behavior, Focus on Past Success was the selected BCT type, and microrandomization resulted in not receiving the message.
Arm/Group | Any Message: Received | Any Message: Not Received | Weighing Message: Received | Weighing Message: Not Received | Weighing BCT 1 Message (Action Planning): Received | Weighing BCT 1 Message (Action Planning): Not Received | Weighing BCT 2 Message (Discrepancy): Received | Weighing BCT 2 Message (Discrepancy): Not Received | Weighing BCT 3 Message (Feedback on Outcome of Behavior): Received | Weighing BCT 3 Message (Feedback on Outcome of Behavior): Not Received | Weighing BCT 4 Message (Social Support): Received | Weighing BCT 4 Message (Social Support): Not Received | Weighing BCT 5 Message (Social Comparison): Received | Weighing BCT 5 Message (Social Comparison): Not Received | Weighing BCT 6 Message (Social Reward): Received | Weighing BCT 6 (Social Reward) Message: Not Received | Weighing BCT 7 Message (Focus on Past Success): Received | Weighing BCT 7 Message (Focus on Past Success): Not Received
Number analyzed (Participants) | 205 | 206 | 205 | 206 | 193 | 194 | 194 | 190 | 196 | 189 | 191 | 195 | 194 | 197 | 0 | 0 | 188 | 191
Number analyzed (Observations) | 25049 | 24935 | 8387 | 8307 | 1401 | 1418 | 1482 | 1400 | 1437 | 1389 | 1436 | 1460 | 1349 | 1333 | 0 | 0 | 1282 | 1307
goals met | 4399 | 4167 | 1496 | 1393 | 249 | 226 | 266 | 247 | 268 | 228 | 237 | 264 | 257 | 210 |  |  | 219 | 218
Statistical Analysis 1: Comparison: Any Message: Received vs Any Message: Not Received; Analysis used generalized estimating equations (GEE) with an independence working residual correlation matrix to account for nesting of observations within individuals. This binary outcome was analyzed using a logit link function. The odds ratio represents the odds of meeting the daily weighing goal among observations in which the participant was randomized to receive a message compared to the odds among observations in which the participant was randomized to not receive a message; Test type: Superiority; p = .03, GEE, logit link function; Odds Ratio (OR) = 1.06, 95% CI 2-sided [1.01 to 1.12]
Statistical Analysis 2: Comparison: Weighing Message: Received vs Weighing Message: Not Received; Analysis used generalized estimating equations (GEE) with an independence working residual correlation matrix to account for nesting of observations within individuals. This binary outcome was analyzed using a logit link function. The odds ratio represents the odds of meeting the daily weighing goal among observations in which the participant was randomized to receive this type of message compared to randomized to not receive this type of message; Test type: Superiority; p = .07, GEE, logit link function; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.99 to 1.17]
Statistical Analysis 3: Comparison: Weighing BCT 1 Message (Action Planning): Received vs Weighing BCT 1 Message (Action Planning): Not Received; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .23, GEE, logit link function; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.92 to 1.41]
Statistical Analysis 4: Comparison: Weighing BCT 2 Message (Discrepancy): Received vs Weighing BCT 2 Message (Discrepancy): Not Received; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .85, GEE, logit link function; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.83 to 1.25]
Statistical Analysis 5: Comparison: Weighing BCT 3 Message (Feedback on Outcome of Behavior): Received vs Weighing BCT 3 Message (Feedback on Outcome of Behavior): Not Received; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .12, GEE, logit link function; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.96 to 1.42]
Statistical Analysis 6: Comparison: Weighing BCT 4 Message (Social Support): Received vs Weighing BCT 4 Message (Social Support): Not Received; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .29, GEE, logit link function; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.74 to 1.09]
Statistical Analysis 7: Comparison: Weighing BCT 5 Message (Social Comparison): Received vs Weighing BCT 5 Message (Social Comparison): Not Received; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .01, GEE, logit link function; Odds Ratio (OR) = 1.26, 95% CI 2-sided [1.05 to 1.51]
Statistical Analysis 8: Comparison: Weighing BCT 7 Message (Focus on Past Success): Received vs Weighing BCT 7 Message (Focus on Past Success): Not Received; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .77, GEE, logit link function; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.84 to 1.25]

2. Primary Outcome: Met Daily Active Minutes Goal
Description: Each observation corresponds to a microrandomization decision point; the reported value reflects the outcome measured within that unit. Among the randomization observations in which the participant had not yet met their active minutes goal, this outcome is the number of observations in which the daily active minutes goal was met after receiving or not receiving a message and before the end of the day. Observations are accumulated across participants and across time. On the day of randomization, a dichotomous outcome of whether a participant met or did not meet their active minutes goal is calculated.
Time Frame: Daily throughout the study, a total of up to 24 weeks
Population: The number of observations analyzed in each arm reflects the total number of observations (across participants, across the study) in which a message of that type was either received or not received, as noted in the arm description. The number of participants analyzed is the total number of participants whose observations are included in that particular arm.
Measure: Number; unit: goals met
Units Other Than Participants: Observations
Groups:
- Active Minutes Message: Received: All observations in which active minutes was the assigned behavior and microrandomization resulted in receiving the message (with any BCT).
- Active Minutes Message: Not Received: All observations in which active minutes was the assigned behavior and microrandomization resulted in not receiving the message (with any BCT).
- Active Minutes BCT 1 Message (Action Planning): Received: All observations in which active minutes was the assigned behavior, Action Planning was the selected BCT type, and microrandomization resulted in receiving the message.
- Active Minutes BCT 1 Message (Action Planning): Not Received: All observations in which active minutes was the assigned behavior, Action Planning was the selected BCT type, and microrandomization resulted in not receiving the message.
- Active Minutes BCT 2 Message (Discrepancy): Received: All observations in which active minutes was the assigned behavior, Discrepancy was the selected BCT type, and microrandomization resulted in receiving the message.
- Active Minutes BCT 2 Message (Discrepancy): Not Received: All observations in which active minutes was the assigned behavior, Discrepancy was the selected BCT type, and microrandomization resulted in not receiving the message.
- Active Minutes BCT 3 Message (Feedback on Outcome of Behavior): Received: All observations in which active minutes was the assigned behavior, Feedback on Outcome of Behavior was the selected BCT type, and microrandomization resulted in receiving the message.
- Active Minutes BCT 3 Message (Feedback on Outcome of Behavior): Not Received: All observations in which active minutes was the assigned behavior, Feedback on Outcome of Behavior was the selected BCT type, and microrandomization resulted in not receiving the message.
- Active Minutes BCT 4 Message (Social Support): Received: All observations in which active minutes was the assigned behavior, Social Support was the selected BCT type, and microrandomization resulted in receiving the message.
- Active Minutes BCT 4 Message (Social Support): Not Received: All observations in which active minutes was the assigned behavior, Social Support was the selected BCT type, and microrandomization resulted in not receiving the message.
- Active Minutes BCT 5 Message (Social Comparison): Received: All observations in which active minutes was the assigned behavior, Social Comparison was the selected BCT type, and microrandomization resulted in receiving the message.
- Active Minutes BCT 5 Message (Social Comparison): Not Received: All observations in which active minutes was the assigned behavior, Social Comparison was the selected BCT type, and microrandomization resulted in not receiving the message.
- Active Minutes BCT 6 Message (Social Reward): Received: All observations in which active minutes was the assigned behavior, Social Reward was the selected BCT type, and microrandomization resulted in receiving the message.
- Active Minutes BCT 6 Message (Social Reward): Not Received: All observations in which active minutes was the assigned behavior, Social Reward was the selected BCT type, and microrandomization resulted in not receiving the message.
- Active Minutes BCT 7 Message (Focus on Past Success): Received: All observations in which active minutes was the assigned behavior, Focus on Past Success was the selected BCT type, and microrandomization resulted in receiving the message.
- Active Minutes BCT 7 Message (Focus on Past Success): Not Received: All observations in which active minutes was the assigned behavior, Focus on Past Success was the selected BCT type, and microrandomization resulted in not receiving the message.
Arm/Group | Any Message: Received | Any Message: Not Received | Active Minutes Message: Received | Active Minutes Message: Not Received | Active Minutes BCT 1 Message (Action Planning): Received | Active Minutes BCT 1 Message (Action Planning): Not Received | Active Minutes BCT 2 Message (Discrepancy): Received | Active Minutes BCT 2 Message (Discrepancy): Not Received | Active Minutes BCT 3 Message (Feedback on Outcome of Behavior): Received | Active Minutes BCT 3 Message (Feedback on Outcome of Behavior): Not Received | Active Minutes BCT 4 Message (Social Support): Received | Active Minutes BCT 4 Message (Social Support): Not Received | Active Minutes BCT 5 Message (Social Comparison): Received | Active Minutes BCT 5 Message (Social Comparison): Not Received | Active Minutes BCT 6 Message (Social Reward): Received | Active Minutes BCT 6 Message (Social Reward): Not Received | Active Minutes BCT 7 Message (Focus on Past Success): Received | Active Minutes BCT 7 Message (Focus on Past Success): Not Received
Number analyzed (Participants) | 206 | 206 | 206 | 206 | 205 | 206 | 206 | 206 | 205 | 206 | 206 | 206 | 205 | 205 | 193 | 194 | 203 | 203
Number analyzed (Observations) | 46097 | 45945 | 15347 | 15353 | 2506 | 2412 | 2336 | 2488 | 2352 | 2378 | 2379 | 2379 | 2324 | 2311 | 1264 | 1253 | 2186 | 2132
goals met | 8781 | 8727 | 2905 | 2959 | 473 | 456 | 410 | 456 | 456 | 474 | 447 | 452 | 397 | 408 | 288 | 292 | 434 | 421
Statistical Analysis 1: Comparison: Any Message: Received vs Any Message: Not Received; Analysis used generalized estimating equations (GEE) with an independence working residual correlation matrix to account for nesting of observations within individuals. This binary outcome was analyzed using a logit link function. The odds ratio represents the odds of meeting the daily active minutes goal among observations in which the participant was randomized to receive a message compared to the odds among observations in which the participant was randomized to not receive a message; Test type: Superiority; p = 1.00, GEE, logit link function; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.97 to 1.04]
Statistical Analysis 2: Comparison: Active Minutes Message: Received vs Active Minutes Message: Not Received; Analysis used generalized estimating equations (GEE) with an independence working residual correlation matrix to account for nesting of observations within individuals. This binary outcome was analyzed using a logit link function. The odds ratio represents the odds of meeting the daily active minutes goal among observations in which the participant was randomized to receive this type of message compared to randomized to not receive this type of message; Test type: Superiority; p = .48, GEE, logit link function; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.92 to 1.03]
Statistical Analysis 3: Comparison: Active Minutes BCT 1 Message (Action Planning): Received vs Active Minutes BCT 1 Message (Action Planning): Not Received; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 1.00, GEE, logit link function; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.85 to 1.17]
Statistical Analysis 4: Comparison: Active Minutes BCT 2 Message (Discrepancy): Received vs Active Minutes BCT 2 Message (Discrepancy): Not Received; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = .48, GEE, logit link function; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.82 to 1.09]
Statistical Analysis 5: Comparison: Active Minutes BCT 3 Message (Feedback on Outcome of Behavior): Received vs Active Minutes BCT 3 Message (Feedback on Outcome of Behavior): Not Received; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = .69, GEE, logit link function; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.83 to 1.12]
Statistical Analysis 6: Comparison: Active Minutes BCT 4 Message (Social Support): Received vs Active Minutes BCT 4 Message (Social Support): Not Received; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = .89, GEE, logit link function; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.85 to 1.14]
Statistical Analysis 7: Comparison: Active Minutes BCT 5 Message (Social Comparison): Received vs Active Minutes BCT 5 Message (Social Comparison): Not Received; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = .61, GEE, logit link function; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.82 to 1.12]
Statistical Analysis 8: Comparison: Active Minutes BCT 6 Message (Social Reward): Received vs Active Minutes BCT 6 Message (Social Reward): Not Received; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = .75, GEE, logit link function; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.81 to 1.17]
Statistical Analysis 9: Comparison: Active Minutes BCT 7 Message (Focus on Past Success): Received vs Active Minutes BCT 7 Message (Focus on Past Success): Not Received; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = .88, GEE, logit link function; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.88 to 1.15]

3. Primary Outcome: At or Under Daily Red Foods Limit
Description: Each observation corresponds to a microrandomization decision point; the reported value reflects the outcome measured within that unit. Among the randomization observations in which the participant had not yet exceeded their red foods limit, this outcome is the number of observations in which the participant stayed at or under their daily red foods limit after receiving or not receiving a message and before the end of the day. Observations are accumulated across participants and across time. On the day of randomization, a dichotomous outcome of whether a participant stayed at or under their red foods limit or did not is calculated.
Time Frame: Daily throughout the study, a total of up to 24 weeks
Population: as for outcome 2
Measure: Number; unit: goals met
Units Other Than Participants: Observations
Groups:
- Red Foods Message: Received: All observations in which red foods was the assigned behavior and microrandomization resulted in receiving the message (with any BCT).
- Red Foods Message: Not Received: All observations in which red foods was the assigned behavior and microrandomization resulted in not receiving the message (with any BCT).
- Red Foods BCT 1 Message (Action Planning): Received: All observations in which red foods was the assigned behavior, Action Planning was the selected BCT type, and microrandomization resulted in receiving the message.
- Red Foods BCT 1 Message (Action Planning): Not Received: All observations in which red foods was the assigned behavior, Action Planning was the selected BCT type, and microrandomization resulted in not receiving the message.
- Red Foods BCT 2 Message (Discrepancy): Received: All observations in which red foods was the assigned behavior, Discrepancy was the selected BCT type, and microrandomization resulted in receiving the message.
- Red Foods BCT 2 Message (Discrepancy): Not Received: All observations in which red foods was the assigned behavior, Discrepancy was the selected BCT type, and microrandomization resulted in not receiving the message.
- Red Foods BCT 3 Message (Feedback on Outcome of Behavior): Received: All observations in which red foods was the assigned behavior, Feedback on Outcome of Behavior was the selected BCT type, and microrandomization resulted in receiving the message.
- Red Foods BCT 3 Message (Feedback on Outcome of Behavior): Not Received: All observations in which red foods was the assigned behavior, Feedback on Outcome of Behavior was the selected BCT type, and microrandomization resulted in not receiving the message.
- Red Foods BCT 4 Message (Social Support): Received: All observations in which red foods was the assigned behavior, Social Support was the selected BCT type, and microrandomization resulted in receiving the message.
- Red Foods BCT 4 Message (Social Support): Not Received: All observations in which red foods was the assigned behavior, Social Support was the selected BCT type, and microrandomization resulted in not receiving the message.
- Red Foods BCT 5 Message (Social Comparison): Received: All observations in which red foods was the assigned behavior, Social Comparison was the selected BCT type, and microrandomization resulted in receiving the message.
- Red Foods BCT 5 Message (Social Comparison): Not Received: All observations in which red foods was the assigned behavior, Social Comparison was the selected BCT type, and microrandomization resulted in not receiving the message.
- Red Foods BCT 6 Message (Social Reward): Received: All observations in which red foods was the assigned behavior, Social Reward was the selected BCT type, and microrandomization resulted in receiving the message.
- Red Foods BCT 6 Message (Social Reward): Not Received: All observations in which red foods was the assigned behavior, Social Reward was the selected BCT type, and microrandomization resulted in not receiving the message.
- Red Foods BCT 7 Message (Focus on Past Success): Received: All observations in which red foods was the assigned behavior, Focus on Past Success was the selected BCT type, and microrandomization resulted in receiving the message.
- Red Foods BCT 7 Message (Focus on Past Success): Not Received: All observations in which red foods was the assigned behavior, Focus on Past Success was the selected BCT type, and microrandomization resulted in not receiving the message.
Arm/Group | Any Message: Received | Any Message: Not Received | Red Foods Message: Received | Red Foods Message: Not Received | Red Foods BCT 1 Message (Action Planning): Received | Red Foods BCT 1 Message (Action Planning): Not Received | Red Foods BCT 2 Message (Discrepancy): Received | Red Foods BCT 2 Message (Discrepancy): Not Received | Red Foods BCT 3 Message (Feedback on Outcome of Behavior): Received | Red Foods BCT 3 Message (Feedback on Outcome of Behavior): Not Received | Red Foods BCT 4 Message (Social Support): Received | Red Foods BCT 4 Message (Social Support): Not Received | Red Foods BCT 5 Message (Social Comparison): Received | Red Foods BCT 5 Message (Social Comparison): Not Received | Red Foods BCT 6 Message (Social Reward): Received | Red Foods BCT 6 Message (Social Reward): Not Received | Red Foods BCT 7 Message (Focus on Past Success): Received | Red Foods BCT 7 Message (Focus on Past Success): Not Received
Number analyzed (Participants) | 206 | 206 | 206 | 206 | 206 | 206 | 205 | 206 | 206 | 206 | 206 | 206 | 206 | 206 | 126 | 141 | 191 | 191
Number analyzed (Observations) | 50335 | 50397 | 16717 | 16896 | 2818 | 2846 | 2760 | 2795 | 2780 | 2818 | 2896 | 2814 | 2686 | 2683 | 440 | 437 | 2337 | 2503
goals met | 13080 | 12848 | 4385 | 4261 | 724 | 711 | 730 | 647 | 715 | 671 | 743 | 708 | 639 | 677 | 201 | 180 | 633 | 667
Statistical Analysis 1: Comparison: Any Message: Received vs Any Message: Not Received; Analysis used generalized estimating equations (GEE) with an independence working residual correlation matrix to account for nesting of observations within individuals. This binary outcome was analyzed using a logit link function. The odds ratio represents the odds of staying at or under the daily red foods limit among observations in which the participant was randomized to receive a message compared to the odds among observations in which the participant was randomized to not receive a message; Test type: Superiority; p = .02, GEE, logit link function; Odds Ratio (OR) = 1.03, 95% CI 2-sided [1.00 to 1.05]
Statistical Analysis 2: Comparison: Red Foods Message: Received vs Red Foods Message: Not Received; Analysis used generalized estimating equations (GEE) with an independence working residual correlation matrix to account for nesting of observations within individuals. This binary outcome was analyzed using a logit link function. The odds ratio represents the odds of staying at or under the daily red foods limit among observations in which the participant was randomized to receive this type of message compared to randomized to not receive this type of message; Test type: Superiority; p = .07, GEE, logit link function; Odds Ratio (OR) = 1.05, 95% CI 2-sided [1.00 to 1.11]
Statistical Analysis 3: Comparison: Red Foods BCT 1 Message (Action Planning): Received vs Red Foods BCT 1 Message (Action Planning): Not Received; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = .49, GEE, logit link function; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.93 to 1.16]
Statistical Analysis 4: Comparison: Red Foods BCT 2 Message (Discrepancy): Received vs Red Foods BCT 2 Message (Discrepancy): Not Received; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = .005, GEE, logit link function; Odds Ratio (OR) = 1.19, 95% CI 2-sided [1.06 to 1.35]
Statistical Analysis 5: Comparison: Red Foods BCT 3 Message (Feedback on Outcome of Behavior): Received vs Red Foods BCT 3 Message (Feedback on Outcome of Behavior): Not Received; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = .09, GEE, logit link function; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.98 to 1.25]
Statistical Analysis 6: Comparison: Red Foods BCT 4 Message (Social Support): Received vs Red Foods BCT 4 Message (Social Support): Not Received; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = .63, GEE, logit link function; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.91 to 1.16]
Statistical Analysis 7: Comparison: Red Foods BCT 5 Message (Social Comparison): Received vs Red Foods BCT 5 Message (Social Comparison): Not Received; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = .17, GEE, logit link function; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.82 to 1.04]
Statistical Analysis 8: Comparison: Red Foods BCT 6 Message (Social Reward): Received vs Red Foods BCT 6 Message (Social Reward): Not Received; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = .20, GEE, logit link function; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.91 to 1.59]
Statistical Analysis 9: Comparison: Red Foods BCT 7 Message (Focus on Past Success): Received vs Red Foods BCT 7 Message (Focus on Past Success): Not Received; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = .74, GEE, logit link function; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.91 to 1.15]

4. Secondary Outcome: Weight Change
Description: Absolute weight change (kg) from baseline to 6 months (6-month weight - baseline weight). Weight was objectively measured on a digital scale in the participant's home.
Time Frame: Baseline, 6 months
Population: This analysis includes the 193 participants who completed the 6-month weight measurement.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Core Behavioral Weight Loss (BWL) Intervention
Number analyzed (Participants) | 193
kg | -2.45 (5.01)
Statistical Analysis 1: Comparison: Core Behavioral Weight Loss (BWL) Intervention; A paired t-test examining change from baseline. (6-month weight - baseline weight); Test type: Superiority; p < .0001, t-test, 2 sided; Mean Difference (Final Values) = -2.45, 95% CI 2-sided [-3.16 to -1.74]

5. Secondary Outcome: Percent Weight Change
Description: Change in weight (%) from baseline to 6 months. Weight will be objectively measured on a digital scale in the participant's home. Percent weight change at 6 months is calculated as ((weight (kg) at 6 months - weight (kg) at baseline)/(weight (kg) at baseline))*100
Time Frame: Baseline, 6 months
Population: This analysis includes only the 193 participants who completed the 6-month weight measurement.
Measure: Mean (Standard Deviation); unit: percent weight change
Arm/Group | Core Behavioral Weight Loss (BWL) Intervention
Number analyzed (Participants) | 193
percent weight change | -2.65 (5.24)
Statistical Analysis 1: Comparison: Core Behavioral Weight Loss (BWL) Intervention; A one-sample t-test evaluating if the mean percent weight change is significantly different than 0. The null hypothesis is that percent weight change is equal to 0; Test type: Superiority; p < .0001, t-test, 2 sided; Mean Difference (Final Values) = -2.65, 95% CI 2-sided [-3.40 to -1.91]

6. Secondary Outcome: Proportion of Days Met Daily Weighing Goal
Description: Calculation of the proportion of study days weighed across all study participants across all days.
Time Frame: Daily throughout the study, a total of up to 24 weeks
Measure: Mean (Standard Deviation); unit: proportion of days
Arm/Group | Core Behavioral Weight Loss (BWL) Intervention
Number analyzed (Participants) | 206
proportion of days | 0.585 (0.280)
Statistical Analysis 1: Comparison: Core Behavioral Weight Loss (BWL) Intervention; A one-sample t-test evaluating if the proportion of days weighed is significantly different from 0; Test type: Superiority; p < .0001, t-test, 2 sided; Mean = 0.585, 95% CI 2-sided [0.547 to 0.624]

7. Secondary Outcome: Proportion of Daily Active Minutes Goal Met
Description: Among randomization observations, the mean proportion of the daily active minutes goal that was achieved that day. Observations are accumulated across participants and across time. Each observation corresponds to a microrandomization decision point; the reported value reflects the outcome measured within that unit. On the day of randomization, a ratio of the participant's total active minutes that day over their daily active minutes goal is calculated (total active minutes that day/daily active minutes goal), such that observations in which a participant exceeded their goal have a proportion over 1.0 and those in which a participant did not reach their active minutes goal have a proportion under 1.0.
Time Frame: Daily throughout the study, a total of up to 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: proportion of active minutes goal met
Units Other Than Participants: Observations
Arm/Group | Any Message: Received | Any Message: Not Received | Active Minutes Message: Received | Active Minutes Message: Not Received | Active Minutes BCT 1 Message (Action Planning): Received | Active Minutes BCT 1 Message (Action Planning): Not Received | Active Minutes BCT 2 Message (Discrepancy): Received | Active Minutes BCT 2 Message (Discrepancy): Not Received | Active Minutes BCT 3 Message (Feedback on Outcome of Behavior): Received | Active Minutes BCT 3 Message (Feedback on Outcome of Behavior): Not Received | Active Minutes BCT 4 Message (Social Support): Received | Active Minutes BCT 4 Message (Social Support): Not Received | Active Minutes BCT 5 Message (Social Comparison): Received | Active Minutes BCT 5 Message (Social Comparison): Not Received | Active Minutes BCT 6 Message (Social Reward): Received | Active Minutes BCT 6 Message (Social Reward): Not Received | Active Minutes BCT 7 Message (Focus on Past Success): Received | Active Minutes BCT 7 Message (Focus on Past Success): Not Received
Number analyzed (Participants) | 206 | 206 | 206 | 206 | 205 | 206 | 206 | 206 | 205 | 206 | 206 | 206 | 205 | 205 | 199 | 195 | 203 | 203
Number analyzed (Observations) | 50986 | 51019 | 16986 | 17003 | 2747 | 2624 | 2547 | 2699 | 2614 | 2644 | 2639 | 2649 | 2529 | 2517 | 1507 | 1519 | 2403 | 2351
proportion of active minutes goal met | 0.795 (1.738) | 0.802 (1.724) | 0.789 (1.705) | 0.808 (1.762) | 0.762 (1.840) | 0.803 (1.985) | 0.739 (1.584) | 0.711 (1.643) | 0.825 (1.732) | 0.863 (1.708) | 0.768 (1.486) | 0.795 (1.519) | 0.689 (1.472) | 0.736 (2.028) | 1.100 (2.246) | 1.063 (1.910) | 0.771 (0.790) | 1.683 (1.504)
Statistical Analysis 1: Comparison: Any Message: Received vs Any Message: Not Received; Analysis used generalized estimating equations (GEE) with an independence working residual correlation matrix to account for nesting of observations within individuals. This ratio outcome was analyzed using a beta link function. The regression coefficient represents the estimated difference in the proportion of the daily active minutes goal that was met among observations in which the participant was randomized to receive a message compared to randomized to not receive a message; Test type: Superiority; p = .43, GEE, beta link function; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.03 to 0.02]
Statistical Analysis 2: Comparison: Active Minutes Message: Received vs Active Minutes Message: Not Received; Analysis used generalized estimating equations (GEE) with an independence working residual correlation matrix to account for nesting of observations within individuals. This ratio outcome was analyzed using a beta link function. The regression coefficient represents the estimated difference in the proportion of the daily active minutes goal that was met among observations in which the participant was randomized to receive this type of message compared to randomized to not receive the message; Test type: Superiority; p = .19, GEE, beta link function; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.05 to 0.01]
Statistical Analysis 3: Comparison: Active Minutes BCT 1 Message (Action Planning): Received vs Active Minutes BCT 1 Message (Action Planning): Not Received; [analysis description as in outcome 7, analysis 2]; Test type: Superiority; p = .50, GEE, beta link function; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.16 to 0.07]
Statistical Analysis 4: Comparison: Active Minutes BCT 2 Message (Discrepancy): Received vs Active Minutes BCT 2 Message (Discrepancy): Not Received; Test type: Superiority; p = .40, GEE, beta link function; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.04 to 0.10]
Statistical Analysis 5: Comparison: Active Minutes BCT 3 Message (Feedback on Outcome of Behavior): Received vs Active Minutes BCT 3 Message (Feedback on Outcome of Behavior): Not Received; [analysis description as in outcome 7, analysis 2]; Test type: Superiority; p = .38, GEE, beta link function; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.13 to 0.05]
Statistical Analysis 6: Comparison: Active Minutes BCT 4 Message (Social Support): Received vs Active Minutes BCT 4 Message (Social Support): Not Received; [analysis description as in outcome 7, analysis 2]; Test type: Superiority; p = .40, GEE, beta link function; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.10 to 0.04]
Statistical Analysis 7: Comparison: Active Minutes BCT 5 Message (Social Comparison): Received vs Active Minutes BCT 5 Message (Social Comparison): Not Received; [analysis description as in outcome 7, analysis 2]; Test type: Superiority; p = .22, GEE, beta link function; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.13 to 0.03]
Statistical Analysis 8: Comparison: Active Minutes BCT 6 Message (Social Reward): Received vs Active Minutes BCT 6 Message (Social Reward): Not Received; [analysis description as in outcome 7, analysis 2]; Test type: Superiority; p = .59, GEE, beta link function; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.11 to 0.18]
Statistical Analysis 9: Comparison: Active Minutes BCT 7 Message (Focus on Past Success): Received vs Active Minutes BCT 7 Message (Focus on Past Success): Not Received; [analysis description as in outcome 7, analysis 2]; Test type: Superiority; p = .62, GEE, beta link function; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.10 to 0.06]

8. Secondary Outcome: Proportion of Daily Red Foods Limit
Description: Among randomization observations, the mean proportion of the daily red foods limit that was tracked that day. Observations are accumulated across participants and across time. Each observation corresponds to a microrandomization decision point; the reported value reflects the outcome measured within that unit. On the day of randomization, a ratio (proportion) of the participant's total red foods that day over their daily red foods limit is calculated (total red foods that day/daily red foods limit), such that observations in which a participant exceeded their limit have a proportion over 1.0 and those in which a participant did not exceed their red foods limit have a proportion under 1.0.
Time Frame: Daily throughout the study, a total of up to 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: proportion of red foods limit
Units Other Than Participants: observations
Arm/Group | Any Message: Received | Any Message: Not Received | Red Foods Message: Received | Red Foods Message: Not Received | Red Foods BCT 1 Message (Action Planning): Received | Red Foods BCT 1 Message (Action Planning): Not Received | Red Foods BCT 2 Message (Discrepancy): Received | Red Foods BCT 2 Message (Discrepancy): Not Received | Red Foods BCT 3 Message (Feedback on Outcome of Behavior): Received | Red Foods BCT 3 Message (Feedback on Outcome of Behavior): Not Received | Red Foods BCT 4 Message (Social Support): Received | Red Foods BCT 4 Message (Social Support): Not Received | Red Foods BCT 5 Message (Social Comparison): Received | Red Foods BCT 5 Message (Social Comparison): Not Received | Red Foods BCT 6 Message (Social Reward): Received | Red Foods BCT 6 Message (Social Reward): Not Received | Red Foods BCT 7 Message (Focus on Past Success): Received | Red Foods BCT 7 Message (Focus on Past Success): Not Received
Number analyzed (Participants) | 197 | 196 | 197 | 194 | 183 | 181 | 178 | 177 | 182 | 179 | 183 | 176 | 169 | 168 | 117 | 125 | 159 | 166
Number analyzed (observations) | 20967 | 20635 | 7001 | 6866 | 1148 | 1129 | 1168 | 1058 | 1147 | 1127 | 1179 | 1140 | 1028 | 1025 | 355 | 341 | 976 | 1046
proportion of red foods limit | 1.042 (0.644) | 1.050 (0.687) | 1.040 (0.644) | 1.052 (0.688) | 1.017 (0.558) | 1.055 (0.670) | 1.043 (0.627) | 1.049 (0.659) | 1.065 (0.764) | 1.088 (0.715) | 1.041 (0.671) | 1.034 (0.661) | 1.014 (0.567) | 1.017 (0.705) | 1.174 (0.760) | 1.171 (0.789) | 1.011 (0.593) | 1.025 (0.677)
Statistical Analysis 1: Comparison: Any Message: Received vs Any Message: Not Received; Analysis used generalized estimating equations (GEE) with an independence working residual correlation matrix to account for nesting of observations within individuals. This ratio outcome was analyzed using a beta link function. The regression coefficient represents the estimated difference in the proportion of the daily red foods limit that was tracked among observations in which the participant was randomized to receive a message compared to randomized to not receive a message; Test type: Superiority; p = 1.00, GEE, beta link function; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.01 to 0.01]
Statistical Analysis 2: Comparison: Red Foods Message: Received vs Red Foods Message: Not Received; Analysis used generalized estimating equations (GEE) with an independence working residual correlation matrix to account for nesting of observations within individuals. This ratio outcome was analyzed using a beta link function. The regression coefficient represents the estimated difference in the proportion of the daily red foods limit that was tracked among observations in which the participant was randomized to receive this type of message compared to randomized to not receive the message; Test type: Superiority; p = .40, GEE, beta link function; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.10 to 0.04]
Statistical Analysis 3: Comparison: Red Foods BCT 1 Message (Action Planning): Received vs Red Foods BCT 1 Message (Action Planning): Not Received; [analysis description as in outcome 8, analysis 2]; Test type: Superiority; p = .38, GEE, beta link function; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.07 to 0.02]
Statistical Analysis 4: Comparison: Red Foods BCT 2 Message (Discrepancy): Received vs Red Foods BCT 2 Message (Discrepancy): Not Received; [analysis description as in outcome 8, analysis 2]; Test type: Superiority; p = 1.00, GEE, beta link function; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.05 to 0.05]
Statistical Analysis 5: Comparison: Red Foods BCT 3 Message (Feedback on Outcome of Behavior): Received vs Red Foods BCT 3 Message (Feedback on Outcome of Behavior): Not Received; [analysis description as in outcome 8, analysis 2]; Test type: Superiority; p = .08, GEE, beta link function; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.09 to 0.00]
Statistical Analysis 6: Comparison: Red Foods BCT 4 Message (Social Support): Received vs Red Foods BCT 4 Message (Social Support): Not Received; [analysis description as in outcome 8, analysis 2]; Test type: Superiority; p = .70, GEE, beta link function; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.04 to 0.06]
Statistical Analysis 7: Comparison: Red Foods BCT 5 Message (Social Comparison): Received vs Red Foods BCT 5 Message (Social Comparison): Not Received; [analysis description as in outcome 8, analysis 2]; Test type: Superiority; p = .33, GEE, beta link function; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.02 to 0.06]
Statistical Analysis 8: Comparison: Red Foods BCT 6 Message (Social Reward): Received vs Red Foods BCT 6 Message (Social Reward): Not Received; [analysis description as in outcome 8, analysis 2]; Test type: Superiority; p = 1.00, GEE, beta link function; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.11 to 0.12]
Statistical Analysis 9: Comparison: Red Foods BCT 7 Message (Focus on Past Success): Received vs Red Foods BCT 7 Message (Focus on Past Success): Not Received; [analysis description as in outcome 8, analysis 2]; Test type: Superiority; p = .70, GEE, beta link function; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.06 to 0.04]

9. Secondary Outcome: Number of Active Minutes
Description: Among randomization observations, the total number of active minutes that was achieved by the participant on the day of randomization. Observations are accumulated across participants and across time. Each observation corresponds to a microrandomization decision point; the reported value reflects the outcome measured within that unit.
Time Frame: Daily throughout the study, a total of up to 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: total active minutes
Units Other Than Participants: observations
Arm/Group | Any Message: Received | Any Message: Not Received | Active Minutes Message: Received | Active Minutes Message: Not Received | Active Minutes BCT 1 Message (Action Planning): Received | Active Minutes BCT 1 Message (Action Planning): Not Received | Active Minutes BCT 2 Message (Discrepancy): Received | Active Minutes BCT 2 Message (Discrepancy): Not Received | Active Minutes BCT 3 Message (Feedback on Outcome of Behavior): Received | Active Minutes BCT 3 Message (Feedback on Outcome of Behavior): Not Received | Active Minutes BCT 4 Message (Social Support): Received | Active Minutes BCT 4 Message (Social Support): Not Received | Active Minutes BCT 5 Message (Social Comparison): Received | Active Minutes BCT 5 Message (Social Comparison): Not Received | Active Minutes BCT 6 Message (Social Reward): Received | Active Minutes BCT 6 Message (Social Reward): Not Received | Active Minutes BCT 7 Message (Focus on Past Success): Received | Active Minutes BCT 7 Message (Focus on Past Success): Not Received
Number analyzed (Participants) | 206 | 206 | 206 | 206 | 205 | 206 | 206 | 206 | 205 | 206 | 206 | 206 | 205 | 205 | 199 | 195 | 203 | 203
Number analyzed (observations) | 50986 | 51019 | 16986 | 17003 | 2747 | 2624 | 2547 | 2699 | 2614 | 2644 | 2639 | 2649 | 2529 | 2517 | 1507 | 1519 | 2403 | 2351
total active minutes | 29.05 (48.33) | 29.44 (48.95) | 28.86 (46.92) | 29.61 (50.29) | 27.36 (44.07) | 28.08 (52.95) | 26.93 (46.93) | 26.96 (49.01) | 28.68 (46.62) | 30.17 (49.80) | 27.92 (44.93) | 28.84 (47.36) | 26.94 (44.50) | 27.80 (51.54) | 39.09 (55.52) | 38.44 (51.61) | 29.43 (48.36) | 30.82 (49.63)
Statistical Analysis 1: Comparison: Any Message: Received vs Any Message: Not Received; Analysis used generalized estimating equations (GEE) with an independence working residual correlation matrix to account for nesting of observations within individuals. The rate ratio reflects the multiplicative change in the number of active minutes per day among observations in which the participant was randomized to receive a message compared to observations in which the participant was randomized to not receive a message; Test type: Superiority; p = .12, GEE, log link function; Rate Ratio = 0.98, 95% CI 2-sided [0.95 to 1.00]
Statistical Analysis 2: Comparison: Active Minutes Message: Received vs Active Minutes Message: Not Received; Analysis used generalized estimating equations (GEE) with an independence working residual correlation matrix to account for nesting of observations within individuals. The rate ratio reflects the multiplicative change in the number of active minutes per day among observations in which the participant was randomized to receive this type of message compared to observations in which the participant was randomized to not receive this type of message; Test type: Superiority; p = .27, GEE, log link function; Rate Ratio = 0.98, 95% CI 2-sided [0.94 to 1.01]
Statistical Analysis 3: Comparison: Active Minutes BCT 1 Message (Action Planning): Received vs Active Minutes BCT 1 Message (Action Planning): Not Received; Test type: Superiority — Analysis used generalized estimating equations (GEE) with an independence working residual correlation matrix to account for nesting of observations within individuals. The rate ratio reflects the multiplicative change in the number of active minutes per day among observations in which the participant was randomized to receive this type of message compared to observations in which the participant was randomized to not receive this type of message; p = .56, GEE, log link function; Rate Ratio = 0.97, 95% CI 2-sided [0.88 to 1.08]
Statistical Analysis 4: Comparison: Active Minutes BCT 2 Message (Discrepancy): Received vs Active Minutes BCT 2 Message (Discrepancy): Not Received; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p = 1.00, GEE, log link function; Rate Ratio = 1.00, 95% CI 2-sided [0.91 to 1.10]
Statistical Analysis 5: Comparison: Active Minutes BCT 3 Message (Feedback on Outcome of Behavior): Received vs Active Minutes BCT 3 Message (Feedback on Outcome of Behavior): Not Received; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p = 0.26, GEE, log link function; Rate Ratio = 0.95, 95% CI 2-sided [0.87 to 1.04]
Statistical Analysis 6: Comparison: Active Minutes BCT 4 Message (Social Support): Received vs Active Minutes BCT 4 Message (Social Support): Not Received; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p = .49, GEE, log link function; Rate Ratio = 0.97, 95% CI 2-sided [0.89 to 1.06]
Statistical Analysis 7: Comparison: Active Minutes BCT 5 Message (Social Comparison): Received vs Active Minutes BCT 5 Message (Social Comparison): Not Received; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p = .54, GEE, log link function; Rate Ratio = 0.97, 95% CI 2-sided [0.88 to 1.07]
Statistical Analysis 8: Comparison: Active Minutes BCT 6 Message (Social Reward): Received vs Active Minutes BCT 6 Message (Social Reward): Not Received; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p = .72, GEE, log link function; Rate Ratio = 1.02, 95% CI 2-sided [0.91 to 1.13]
Statistical Analysis 9: Comparison: Active Minutes BCT 7 Message (Focus on Past Success): Received vs Active Minutes BCT 7 Message (Focus on Past Success): Not Received; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p = .34, GEE, log link function; Rate Ratio = 0.96, 95% CI 2-sided [0.88 to 1.04]

10. Secondary Outcome: Number of Red Foods
Description: Among randomization observations, the total number of red foods that was tracked by the participant on the day of randomization. Observations are accumulated across participants and across time. Each observation corresponds to a microrandomization decision point; the reported value reflects the outcome measured within that unit.
Time Frame: Daily throughout the study, a total of up to 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: total red foods
Units Other Than Participants: Observations
Arm/Group | Any Message: Received | Any Message: Not Received | Red Foods Message: Received | Red Foods Message: Not Received | Red Foods BCT 1 Message (Action Planning): Received | Red Foods BCT 1 Message (Action Planning): Not Received | Red Foods BCT 2 Message (Discrepancy): Received | Red Foods BCT 2 Message (Discrepancy): Not Received | Red Foods BCT 3 Message (Feedback on Outcome of Behavior): Received | Red Foods BCT 3 Message (Feedback on Outcome of Behavior): Not Received | Red Foods BCT 4 Message (Social Support): Received | Red Foods BCT 4 Message (Social Support): Not Received | Red Foods BCT 5 Message (Social Comparison): Received | Red Foods BCT 5 Message (Social Comparison): Not Received | Red Foods BCT 6 Message (Social Reward): Received | Red Foods BCT 6 Message (Social Reward): Not Received | Red Foods BCT 7 Message (Focus on Past Success): Received | Red Foods BCT 7 Message (Focus on Past Success): Not Received
Number analyzed (Participants) | 197 | 196 | 197 | 194 | 183 | 181 | 178 | 177 | 182 | 179 | 183 | 176 | 169 | 168 | 117 | 125 | 159 | 166
Number analyzed (Observations) | 20967 | 20635 | 7001 | 6866 | 1148 | 1129 | 1168 | 1058 | 1147 | 1127 | 1179 | 1140 | 1028 | 1025 | 355 | 341 | 976 | 1046
total red foods | 3.45 (2.08) | 3.47 (2.14) | 3.45 (2.08) | 3.47 (2.14) | 3.39 (1.96) | 3.48 (2.07) | 3.48 (2.04) | 3.47 (2.03) | 3.49 (2.20) | 3.61 (2.29) | 3.44 (2.16) | 3.45 (2.16) | 3.39 (1.99) | 3.32 (2.08) | 3.79 (2.18) | 3.79 (2.30) | 3.37 (2.03) | 3.39 (2.14)
Statistical Analysis 1: Comparison: Any Message: Received vs Any Message: Not Received; Analysis used generalized estimating equations (GEE) with an independence working residual correlation matrix to account for nesting of observations within individuals. The rate ratio reflects the multiplicative change in the number of red foods day among observations in which the participant was randomized to receive a message compared to observations in which the participant was randomized to not receive a message; Test type: Superiority; p = 1.00, GEE, log link function; Rate Ratio = 1.00, 95% CI 2-sided [0.98 to 1.01]
Statistical Analysis 2: Comparison: Red Foods Message: Received vs Red Foods Message: Not Received; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = .33, GEE, log link function; Rate Ratio = 0.99, 95% CI 2-sided [0.97 to 1.01]
Statistical Analysis 3: Comparison: Red Foods BCT 1 Message (Action Planning): Received vs Red Foods BCT 1 Message (Action Planning): Not Received; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = .20, GEE, log link function; Rate Ratio = 0.97, 95% CI 2-sided [0.93 to 1.02]
Statistical Analysis 4: Comparison: Red Foods BCT 2 Message (Discrepancy): Received vs Red Foods BCT 2 Message (Discrepancy): Not Received; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 1.00, GEE, log link function; Rate Ratio = 1.00, 95% CI 2-sided [0.95 to 1.05]
Statistical Analysis 5: Comparison: Red Foods BCT 3 Message (Feedback on Outcome of Behavior): Received vs Red Foods BCT 3 Message (Feedback on Outcome of Behavior): Not Received; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = .09, GEE, log link function; Rate Ratio = 0.96, 95% CI 2-sided [0.92 to 1.01]
Statistical Analysis 6: Comparison: Red Foods BCT 4 Message (Social Support): Received vs Red Foods BCT 4 Message (Social Support): Not Received; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = .63, GEE, log link function; Rate Ratio = 1.03, 95% CI 2-sided [0.91 to 1.16]
Statistical Analysis 7: Comparison: Red Foods BCT 5 Message (Social Comparison): Received vs Red Foods BCT 5 Message (Social Comparison): Not Received; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = .17, GEE, log link function; Rate Ratio = 0.92, 95% CI 2-sided [0.82 to 1.04]
Statistical Analysis 8: Comparison: Red Foods BCT 6 Message (Social Reward): Received vs Red Foods BCT 6 Message (Social Reward): Not Received; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = .20, GEE, log link function; Rate Ratio = 1.20, 95% CI 2-sided [0.91 to 1.59]
Statistical Analysis 9: Comparison: Red Foods BCT 7 Message (Focus on Past Success): Received vs Red Foods BCT 7 Message (Focus on Past Success): Not Received; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = .74, GEE, log link function; Rate Ratio = 1.02, 95% CI 2-sided [0.91 to 1.15]

11. Secondary Outcome: Met Daily Weighing Goal Tomorrow
Description: Each observation corresponds to a microrandomization decision point; the reported value reflects the outcome measured within that unit. Among the randomization observations, this outcome is the number of observations in which the daily weighing goal was met the day following randomization. Observations are accumulated across participants and across time. On the day following randomization, a dichotomous outcome of whether a participant weighed or did not weigh is assessed.
Time Frame: Daily throughout the study, a total of up to 24 weeks
Population: as for outcome 2
Measure: Number; unit: goals met
Units Other Than Participants: Observations
Groups:
- Weighing BCT 6 Message (Social Reward): Not Received: All observations in which weighing was the assigned behavior, Social Reward was the selected BCT type, and microrandomization resulted in not receiving the message.
Arm/Group | Any Message: Received | Any Message: Not Received | Weighing Message: Received | Weighing Message: Not Received | Weighing BCT 1 Message (Action Planning): Received | Weighing BCT 1 Message (Action Planning): Not Received | Weighing BCT 2 Message (Discrepancy): Received | Weighing BCT 2 Message (Discrepancy): Not Received | Weighing BCT 3 Message (Feedback on Outcome of Behavior): Received | Weighing BCT 3 Message (Feedback on Outcome of Behavior): Not Received | Weighing BCT 4 Message (Social Support): Received | Weighing BCT 4 Message (Social Support): Not Received | Weighing BCT 5 Message (Social Comparison): Received | Weighing BCT 5 Message (Social Comparison): Not Received | Weighing BCT 6 Message (Social Reward): Received | Weighing BCT 6 Message (Social Reward): Not Received | Weighing BCT 7 Message (Focus on Past Success): Received | Weighing BCT 7 Message (Focus on Past Success): Not Received
Number analyzed (Participants) | 206 | 206 | 206 | 206 | 205 | 205 | 194 | 190 | 206 | 205 | 206 | 206 | 206 | 205 | 195 | 197 | 203 | 203
Number analyzed (Observations) | 50986 | 51019 | 17079 | 16924 | 2823 | 2883 | 1482 | 1400 | 2937 | 2878 | 2999 | 2901 | 2719 | 2682 | 1425 | 1514 | 2694 | 2666
goals met | 29985 | 29969 | 10022 | 9959 | 1637 | 1682 | 487 | 461 | 1751 | 1723 | 1781 | 1744 | 1581 | 1527 | 1189 | 1246 | 1596 | 1576
Statistical Analysis 1: Comparison: Any Message: Received vs Any Message: Not Received; Analysis used generalized estimating equations (GEE) with an independence working residual correlation matrix to account for nesting of observations within individuals. This binary outcome was analyzed using a logit link function. The odds ratio represents the odds of meeting the daily weighing goal the following day among observations in which the participant was randomized to receive a message compared to randomized to not receive a message; Test type: Superiority; p = 1.00, GEE, logit link function; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.98 to 1.03]
Statistical Analysis 2: Comparison: Weighing Message: Received vs Weighing Message: Not Received; Analysis used generalized estimating equations (GEE) with an independence working residual correlation matrix to account for nesting of observations within individuals. This binary outcome was analyzed using a logit link function. The odds ratio represents the odds of meeting the daily weighing goal the following day among observations in which the participant was randomized to receive this type of message compared to randomized to not receive this type of message; Test type: Superiority; p = .66, GEE, logit link function; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.95 to 1.04]
Statistical Analysis 3: Comparison: Weighing BCT 1 Message (Action Planning): Received vs Weighing BCT 1 Message (Action Planning): Not Received; [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p = .74, GEE, logit link function; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.87 to 1.10]
Statistical Analysis 4: Comparison: Weighing BCT 2 Message (Discrepancy): Received vs Weighing BCT 2 Message (Discrepancy): Not Received; [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p = 1.00, GEE, logit link function; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.86 to 1.16]
Statistical Analysis 5: Comparison: Weighing BCT 3 Message (Feedback on Outcome of Behavior): Received vs Weighing BCT 3 Message (Feedback on Outcome of Behavior): Not Received; [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p = .84, GEE, logit link function; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.90 to 1.09]
Statistical Analysis 6: Comparison: Weighing BCT 4 Message (Social Support): Received vs Weighing BCT 4 Message (Social Support): Not Received; [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p = .39, GEE, logit link function; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.88 to 1.06]
Statistical Analysis 7: Comparison: Weighing BCT 5 Message (Social Comparison): Received vs Weighing BCT 5 Message (Social Comparison): Not Received; [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p = .36, GEE, logit link function; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.95 to 1.17]
Statistical Analysis 8: Comparison: Weighing BCT 6 Message (Social Reward): Received vs Weighing BCT 6 Message (Social Reward): Not Received; [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p = .44, GEE, logit link function; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.89 to 1.31]
Statistical Analysis 9: Comparison: Weighing BCT 7 Message (Focus on Past Success): Received vs Weighing BCT 7 Message (Focus on Past Success): Not Received; [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p = .86, GEE, logit link function; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.90 to 1.13]

12. Secondary Outcome: Met Daily Active Minutes Goal Tomorrow
Description: Each observation corresponds to a microrandomization decision point; the reported value reflects the outcome measured within that unit. Among the randomization observations, this outcome is the number of observations in which the daily active minutes goal was met the day following randomization. Observations are accumulated across participants and across time. On the day following randomization, a dichotomous outcome of whether a participant met or did not meet their active minutes goal is calculated.
Time Frame: Daily throughout the study, a total of up to 24 weeks
Population: as for outcome 2
Measure: Number; unit: goals met
Units Other Than Participants: Observations
Arm/Group | Any Message: Received | Any Message: Not Received | Active Minutes Message: Received | Active Minutes Message: Not Received | Active Minutes BCT 1 Message (Action Planning): Received | Active Minutes BCT 1 Message (Action Planning): Not Received | Active Minutes BCT 2 Message (Discrepancy): Received | Active Minutes BCT 2 Message (Discrepancy): Not Received | Active Minutes BCT 3 Message (Feedback on Outcome of Behavior): Received | Active Minutes BCT 3 Message (Feedback on Outcome of Behavior): Not Received | Active Minutes BCT 4 Message (Social Support): Received | Active Minutes BCT 4 Message (Social Support): Not Received | Active Minutes BCT 5 Message (Social Comparison): Received | Active Minutes BCT 5 Message (Social Comparison): Not Received | Active Minutes BCT 6 Message (Social Reward): Received | Active Minutes BCT 6 Message (Social Reward): Not Received | Active Minutes BCT 7 Message (Focus on Past Success): Received | Active Minutes BCT 7 Message (Focus on Past Success): Not Received
Number analyzed (Participants) | 206 | 206 | 206 | 206 | 205 | 206 | 206 | 206 | 205 | 206 | 206 | 206 | 205 | 205 | 199 | 195 | 203 | 203
Number analyzed (Observations) | 50986 | 51019 | 16986 | 17003 | 2747 | 2624 | 2547 | 2699 | 2614 | 2644 | 2639 | 2649 | 2529 | 2517 | 1507 | 1519 | 2403 | 2351
goals met | 13415 | 13472 | 4452 | 4501 | 709 | 670 | 650 | 639 | 647 | 718 | 701 | 722 | 617 | 601 | 505 | 509 | 623 | 642
Statistical Analysis 1: Comparison: Any Message: Received vs Any Message: Not Received; Analysis used generalized estimating equations (GEE) with an independence working residual correlation matrix to account for nesting of observations within individuals. This binary outcome was analyzed using a logit link function. The odds ratio represents the odds of meeting the daily active minutes goal the following day among observations in which the participant was randomized to receive a message compared to randomized to not receive a message; Test type: Superiority; p = 1.00, GEE, logit link function; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.97 to 1.02]
Statistical Analysis 2: Comparison: Any Message: Not Received vs Active Minutes Message: Received; Analysis used generalized estimating equations (GEE) with an independence working residual correlation matrix to account for nesting of observations within individuals. This binary outcome was analyzed using a logit link function. The odds ratio represents the odds of meeting the daily active minutes goal the following day among observations in which the participant was randomized to receive this type of message compared to randomized to not receive this type of message; Test type: Superiority; p = .67, GEE, logit link function; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.94 to 1.03]
Statistical Analysis 3: Comparison: Active Minutes BCT 1 Message (Action Planning): Received vs Active Minutes BCT 1 Message (Action Planning): Not Received; [analysis description as in outcome 12, analysis 2]; Test type: Superiority; p = .82, GEE, logit link function; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.93 to 1.10]
Statistical Analysis 4: Comparison: Active Minutes BCT 2 Message (Discrepancy): Received vs Active Minutes BCT 2 Message (Discrepancy): Not Received; [analysis description as in outcome 12, analysis 2]; Test type: Superiority; p = .09, GEE, logit link function; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.99 to 1.18]
Statistical Analysis 5: Comparison: Active Minutes BCT 3 Message (Feedback on Outcome of Behavior): Received vs Active Minutes BCT 3 Message (Feedback on Outcome of Behavior): Not Received; [analysis description as in outcome 12, analysis 2]; Test type: Superiority; p = .05, GEE, logit link function; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.83 to 1.00]
Statistical Analysis 6: Comparison: Active Minutes BCT 4 Message (Social Support): Received vs Active Minutes BCT 4 Message (Social Support): Not Received; [analysis description as in outcome 12, analysis 2]; Test type: Superiority; p = .63, GEE, logit link function; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.90 to 1.06]
Statistical Analysis 7: Comparison: Active Minutes BCT 5 Message (Social Comparison): Received vs Active Minutes BCT 5 Message (Social Comparison): Not Received; [analysis description as in outcome 12, analysis 2]; Test type: Superiority; p = .69, GEE, logit link function; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.93 to 1.13]
Statistical Analysis 8: Comparison: Active Minutes BCT 6 Message (Social Reward): Received vs Active Minutes BCT 6 Message (Social Reward): Not Received; [analysis description as in outcome 12, analysis 2]; Test type: Superiority; p = 1.00, GEE, logit link function; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.91 to 1.10]
Statistical Analysis 9: Comparison: Active Minutes BCT 7 Message (Focus on Past Success): Received vs Active Minutes BCT 7 Message (Focus on Past Success): Not Received; [analysis description as in outcome 12, analysis 2]; Test type: Superiority; p = .31, GEE, logit link function; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.86 to 1.05]

13. Secondary Outcome: At or Under Daily Red Foods Limit Tomorrow
Description: Each observation corresponds to a microrandomization decision point; the reported value reflects the outcome measured within that unit. Among the randomization observations, this outcome is the number of observations in which the participant stayed at or under the daily red foods limit the day following randomization. Observations are accumulated across participants and across time. On the day following randomization, a dichotomous outcome of whether a participant stayed at or under the daily red foods limit is calculated.
Time Frame: Daily throughout the study, a total of up to 24 weeks
Population: as for outcome 2
Measure: Number; unit: goals met
Units Other Than Participants: Observations
Arm/Group | Any Message: Received | Any Message: Not Received | Red Foods Message: Received | Red Foods Message: Not Received | Red Foods BCT 1 Message (Action Planning): Received | Red Foods BCT 1 Message (Action Planning): Not Received | Red Foods BCT 2 Message (Discrepancy): Received | Red Foods BCT 2 Message (Discrepancy): Not Received | Red Foods BCT 3 Message (Feedback on Outcome of Behavior): Received | Red Foods BCT 3 Message (Feedback on Outcome of Behavior): Not Received | Red Foods BCT 4 Message (Social Support): Received | Red Foods BCT 4 Message (Social Support): Not Received | Red Foods BCT 5 Message (Social Comparison): Received | Red Foods BCT 5 Message (Social Comparison): Not Received | Red Foods BCT 6 Message (Social Reward): Received | Red Foods BCT 6 Message (Social Reward): Not Received | Red Foods BCT 7 Message (Focus on Past Success): Received | Red Foods BCT 7 Message (Focus on Past Success): Not Received
Number analyzed (Participants) | 206 | 206 | 206 | 206 | 206 | 206 | 205 | 206 | 206 | 206 | 206 | 206 | 206 | 206 | 133 | 145 | 191 | 191
Number analyzed (Observations) | 50986 | 51019 | 16921 | 17092 | 2846 | 2868 | 2789 | 2826 | 2815 | 2852 | 2923 | 2848 | 2715 | 2706 | 482 | 472 | 2351 | 2520
goals met | 12875 | 12793 | 4245 | 4312 | 680 | 674 | 703 | 688 | 700 | 709 | 726 | 697 | 606 | 672 | 207 | 196 | 623 | 676
Statistical Analysis 1: Comparison: Any Message: Received vs Any Message: Not Received; Analysis used generalized estimating equations (GEE) with an independence working residual correlation matrix to account for nesting of observations within individuals. This binary outcome was analyzed using a logit link function. The odds ratio represents the odds of staying at or under the daily red foods limit the following day among observations in which the participant was randomized to receive a message compared to randomized to not receive a message; Test type: Superiority; p = .51, GEE, logit link function; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.98 to 1.04]
Statistical Analysis 2: Comparison: Red Foods Message: Received vs Red Foods Message: Not Received; Analysis used generalized estimating equations (GEE) with an independence working residual correlation matrix to account for nesting of observations within individuals. This binary outcome was analyzed using a logit link function. The odds ratio represents the odds of staying at or under the daily red foods limit the following day among observations in which the participant was randomized to receive this type of message compared to randomized to not receive this type of message; Test type: Superiority; p = .70, GEE, logit link function; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.94 to 1.04]
Statistical Analysis 3: Comparison: Red Foods BCT 1 Message (Action Planning): Received vs Red Foods BCT 1 Message (Action Planning): Not Received; [analysis description as in outcome 13, analysis 2]; Test type: Superiority; p = .76, GEE, logit link function; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.90 to 1.16]
Statistical Analysis 4: Comparison: Red Foods BCT 2 Message (Discrepancy): Received vs Red Foods BCT 2 Message (Discrepancy): Not Received; [analysis description as in outcome 13, analysis 2]; Test type: Superiority; p = .38, GEE, logit link function; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.94 to 1.17]
Statistical Analysis 5: Comparison: Red Foods BCT 3 Message (Feedback on Outcome of Behavior): Received vs Red Foods BCT 3 Message (Feedback on Outcome of Behavior): Not Received; [analysis description as in outcome 13, analysis 2]; Test type: Superiority; p = .87, GEE, logit link function; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.88 to 1.13]
Statistical Analysis 6: Comparison: Red Foods BCT 4 Message (Social Support): Received vs Red Foods BCT 4 Message (Social Support): Not Received; [analysis description as in outcome 13, analysis 2]; Test type: Superiority; p = .74, GEE, logit link function; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.90 to 1.14]
Statistical Analysis 7: Comparison: Red Foods BCT 5 Message (Social Comparison): Received vs Red Foods BCT 5 Message (Social Comparison): Not Received; [analysis description as in outcome 13, analysis 2]; Test type: Superiority; p = .03, GEE, logit link function; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.76 to 0.99]
Statistical Analysis 8: Comparison: Red Foods BCT 6 Message (Social Reward): Received vs Red Foods BCT 6 Message (Social Reward): Not Received; [analysis description as in outcome 13, analysis 2]; Test type: Superiority; p = .66, GEE, logit link function; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.82 to 1.38]
Statistical Analysis 9: Comparison: Red Foods BCT 7 Message (Focus on Past Success): Received vs Red Foods BCT 7 Message (Focus on Past Success): Not Received; [analysis description as in outcome 13, analysis 2]; Test type: Superiority; p = .75, GEE, logit link function; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.87 to 1.11]

ADVERSE EVENTS:
Time Frame: up to 6 months
Arm/Group | Core Behavioral Weight Loss (BWL) Intervention
All-Cause Mortality (participants affected / at risk) | 0/206
Serious Adverse Events (participants affected / at risk) | 0/206
Other Adverse Events (participants affected / at risk) | 12/206
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Core Behavioral Weight Loss (BWL) Intervention (N=206)
Ankle sprain (Injury, poisoning and procedural complications) | 4
Muscle strain (Musculoskeletal and connective tissue disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-12): https://cdn.clinicaltrials.gov/large-docs/61/NCT05625061/Prot_SAP_001.pdf
  • Informed Consent Form (2023-12-12): https://cdn.clinicaltrials.gov/large-docs/61/NCT05625061/ICF_000.pdf